CLINICAL TRIAL: NCT04890535
Title: Phase 1, Partially Blinded, Placebo-Controlled, Randomized, Combined Single Ascending Dose With Food Effect Cohort Trial and Multiple Ascending Dose Trial to Evaluate the Safety, Tolerability, and PK of TBAJ-587 in Healthy Adults
Brief Title: Evaluation of the Safety, Tolerability, PK of TBAJ-587 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Global Alliance for TB Drug Development (Other)
Collaborators: QPS Holdings LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TBAJ-587-CL001
Record Dates: First submitted 2021-02-19; First posted 2021-05-18 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Tuberculosis
Keywords: Phase I
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Single Ascending Dose 25 - 800 mg (Active Comparator): single dose of TBAJ-587
  Interventions: Drug: TBAJ-587
- Single Ascending Dose 25 - 800 mg placebo (Placebo Comparator): single dose of placebo
  Interventions: Drug: Placebo
- Multiple Ascending Dose 50 - 200 mg (Active Comparator): 28 days dose of TBAJ-587
  Interventions: Drug: TBAJ-587
- Multiple Ascending Dose 50 - 200 mg Placebo (Placebo Comparator): 28 days dose of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TBAJ-587 — oral suspension
  Arms: Multiple Ascending Dose 50 - 200 mg; Single Ascending Dose 25 - 800 mg
Drug: Placebo — matching placebo oral suspension for TBAJ-587
  Arms: Multiple Ascending Dose 50 - 200 mg Placebo; Single Ascending Dose 25 - 800 mg placebo

SUMMARY:
Phase 1, Partially Blinded, Placebo-Controlled, Randomized, Combined Single Ascending Dose with Food Effect Cohort Trial (Part 1) and Multiple Ascending Dose Trial (Part 2) to Evaluate the Safety, Tolerability, and PK of TBAJ-587 in Healthy Adults

DETAILED DESCRIPTION:
This is a two-part, partially blinded, placebo-controlled, combined single ascending dose (SAD) trial with a food-effect cohort (Part 1) and multiple ascending dose (MAD) trial (Part 2) to be conducted in one trial centre in Europe.

Part 1: Has a single ascending dose (SAD) design with up to 6 planned dose levels with a food-effect cohort at one of the dose levels.

The first SAD cohort will be separated into 2 groups. A sentinel group of two participants (1 active and 1 placebo) will be dosed at least 72 hours before the remaining 6 participants (5 active and 1 placebo). The other cohorts will not be separated.

Other Dose Level cohorts: scheduling of safety and PK sample collection will be based on the PK data collected from previous cohorts.

Food-Effect Cohort: Based on exposure levels from preceding SAD cohorts, one of the planned cohorts and the specific dose will be selected for the food effect (FE) cohort which will study the effect on PK after a high-calorie, high-fat meal. Additional participants will be recruited to reach a total of 9 active participants, inclusive of the previously dosed participants, in the fasted group, and 9 additional active participants will be recruited for the group dosed with food.

Note: The decision to proceed to the next cohort will be based on a Dose Escalation Meeting (DEM) which will take place after the Day 7 PK profile and approximately 14 days of safety data is available depending on the time required for PK analysis. The EC will be notified on the outcome of the DEM and the next cohort will start once the EC grants approval. The scheduling and duration of the PK and safety data collection for the DEM may be revised based on what is learned about the PK and safety from the initial cohorts during Part 1 of the trial. This PK and safety data might also impact the scheduling of the PK collection/sampling and safety assessments for the remainder of the cohorts in Part 1 and Part 2.

Participants will continue to be monitored for safety which may continue up to approximately 20 weeks after the last dose if indicated by interim PK analysis.

At the end of Part 1 (SAD), pharmacokinetic and safety data along with rationale for choosing the doses for the multiple ascending dose (MAD) part, Part 2, will be submitted to the Ethics Committee (EC). The trial will not proceed to Part 2 until the Sponsor, in conjunction with the Principal Investigator (PI) and members of the Safety Review Committee (SRC) at the DEM, has determined that adequate safety, tolerability, and PKs from the Part 1 cohorts have been demonstrated and all required parties, including the EC, have provided approval.

Part 2: Has a multiple ascending dose (MAD) design. Three cohorts are planned for Part 2 and will be determined based on model predictions of steady state AUC exposures and safety from Part 1.

In this MAD part, each participant, based on current assumptions, is expected to be administered TBAJ-587 or matching placebo daily for 28 days with corresponding PK and safety measurements.

Note: The DEM will be scheduled after the Day 14 PK profile data is available depending on the time required for PK analysis. The EC will be notified, and the next cohort will start once the EC grants approval.

The safety and PK collection/sampling schedule for the MAD may be revised based on what is learned about the PK and safety from Part 1 of the trial. Furthermore, with regard to the DEM, the timing and duration of the safety and PK sampling needed to decide on escalating to the next dose will also be determined and finalized based on the PK data obtained from Part 1.

Participants will continue to be monitored for safety at time points up to approximately 20 weeks after the last dose if indicated by interim PK analysis.

Additional cohorts: up to three additional cohorts in Part 1 and one additional cohort in Part 2 may be enrolled if deemed appropriate by the Sponsor to repeat a dose level or to study another dose level.

Dose escalation to the next cohort (i.e. next dose level), the decision for the trial to progress to the planned MAD cohorts (Part 2), any changes to the PK sampling and safety assessment time points, or the decisions on additional cohorts will not take place until the Sponsor, in conjunction with the PI and members of the SRC at the DEM, has determined that adequate safety, tolerability, and pharmacokinetics from the previous cohort have been demonstrated to permit proceeding to the next cohort. The EC should be notified, and the decision can only be implemented once the EC grants approval.

Interim PK analyses (the prediction PK model may be modified if necessary) and safety assessments will be performed for the dose escalation decisions, to select the intermediate dose for the food effect cohort, and to reconsider (if needed) the sampling time points as the trial progresses. All samples will be sent for analysis and the bioanalytical lab will be unblinded and run the analysis on active treatment participants only. Data from the analysis used for the dose escalation meetings will only include active treatment participants and will be blinded by participant for the Sponsor trial team, PI and SRC members.

Safety will be assessed throughout the trial. Physical examinations, safety laboratory, vital signs, serial Electrocardiograms (ECGs), Holter monitoring and serial blood samples will be collected for safety and PK assessment of TBAJ-587 and metabolites.

As data from each cohort is informative for dose escalation decisions in subsequent cohorts, review of unblinded data will be conducted by 2 experienced individuals not directly involved in the study, one of whom must be a physician. Upon completion of the review, they will communicate to the study team and SRC modifications, if any, that should be implemented for subsequent cohorts.

ELIGIBILITY:
Inclusion Criteria:

Participants are required to meet all the following inclusion criteria to be eligible for participation in the trial:

1. Provide written, informed consent prior to all trial-related procedures.
2. Healthy adult male and females of non-childbearing potential, 18-64 years of age (inclusive) at the time of screening.
3. Body mass index (BMI) ≥ 18.5 and ≤ 32.0 (kg/m2) and a body weight of no less than 50.0 kg.
4. Medically healthy with no clinically significant screening results (e.g., laboratory profiles normal or up to Grade 1 per FDA Toxicity Grading Scale), medical histories, vital signs, ECGs, physical examination findings, as deemed by the Investigator. Lab results within the testing facilities normal range will not be considered AEs when referenced to the FDA (Appendix 2) assessment/grading scale. If exclusionary lab criteria are met, values may be confirmed by repeat evaluation.
5. No use of tobacco or nicotine containing products (including smoking cessation products), for a minimum of 6 months prior to dosing.
6. Females of non-childbearing potential, having undergone one of the following sterilization procedures at least 6 months prior to dosing:

   1. Hysteroscopic sterilization
   2. Bilateral tubal ligation or bilateral salpingectomy
   3. Hysterectomy
   4. Bilateral oophorectomy or be postmenopausal with amenorrhea for at least 1 year prior to the first dose with serum
   5. Follicle-stimulating hormone (FSH) levels consistent with postmenopausal status at screening.
7. Non-vasectomized males (or males vasectomized less than 120 days prior to trial start), must agree to the following during trial participation and for 90 days following the last administration of trial drug:

   1. Use a condom with spermicide while engaging in sexual activity or be sexually abstinent
   2. Not donate sperm during this time.
8. In the event the sexual partner is surgically sterile, use of a condom with spermicide is not necessary.
9. None of the restrictions listed above are required for vasectomized males whose procedure was performed more than 120 days prior to trial start.
10. Willing to answer inclusion and exclusion criteria questionnaire at check-in.
11. Participant understands trial procedures and provides written informed consent for the trial.
12. Be able to comply with the protocol and the assessments therein, including all restrictions.
13. Is willing and able to remain in the trial unit for the entire duration of the assigned confinement period and return for outpatient visits.
14. If enrolled in Part 1 and assigned to the fasted/fed cohort, is willing and able to consume the entire high-calorie, high-fat breakfast meal in the timeframe required.
15. Has negative Quantiferon test during the screening. -

Exclusion Criteria:

Participants will be excluded from the trial if there is evidence of any of the following criteria at screening or check-in, as appropriate.

1. History or presence of significant cardiovascular abnormalities, Heart Murmur, pulmonary, hepatic, renal, haematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease as determined by the Investigator to be clinically relevant.
2. Any musculoskeletal abnormality (severe tenderness with marked impairment of activity) or musculoskeletal toxicity (frank necrosis).
3. History of any illness that, in the opinion of the Investigator, might confound the results of the trial or poses an additional risk to the participant by their participation in the trial.
4. Surgery within the past 90 days prior to dosing or other previous surgery as determined by the Investigator to be clinically relevant.
5. History or presence of alcoholism or drug abuse within the past 2 years as determined by the Investigator to be clinically relevant.
6. Female participants who are pregnant or lactating.
7. Positive results for the urine drug/alcohol breath screen at screening or check-in.
8. Positive urine cotinine at screening or check-in.
9. Participants with the following laboratory abnormalities at screening:

   1. ALT or AST >1.0 times ULN
   2. Creatinine grade 2 or greater (>1.5 times ULN)
   3. Total lipase or amylase >1.0 times ULN
   4. Total bilirubin grade 1 or greater (>1.0 times ULN)
   5. CPK >1.25 times ULN If exclusionary lab criteria are met, values may be confirmed by repeat evaluation.
10. Positive results at screening for Human Immunodeficiency Virus (HIV), Hepatitis B Surface Antigen (HBsAg), or Hepatitis C antibodies (HCV).
11. Positive severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) results at screening.
12. Seated or supine blood pressure is less than 90/40 mmHg or greater than 150/90 mmHg at screening, Day -2 (check-in), Day -1, or pre-dose. Out of range vital signs may be repeated once for confirmation.

    Out of range values will not be considered AEs if the repeat assessment is in range.
13. Heart rate is lower than 40 bpm or higher than 100 bpm at screening, Day -2 (check-in), Day -1, or pre-dose. Out of range vital signs may be repeated once for confirmation. Out of range values will not be considered AE s if the repeat assessment is in range.
14. Any clinically significant electrocardiogram abnormality at Screening (as deemed by decision of the Investigator and the Sponsor's Medical Monitor).

    NOTE: The following can be considered not clinically significant without consulting the Sponsor's Medical Monitor:
    1. Mild first-degree A-V block (P-R interval <0.23 sec)
    2. Right or left axis deviation
    3. Incomplete right bundle branch block
    4. Isolated left anterior fascicular block (left anterior hemiblock) in younger athletic participants
15. QTcF interval >450 ms for males or >470 ms for females at screening, Day -2, Day -1, or Day 1 (pre-dose), or history of prolonged QT syndrome. For triplicate ECGs taken at screening and Day-2, the average QTcF interval of the three ECG recordings will be used to determine qualification.
16. Family history of Long-QT Syndrome or sudden death without a preceding diagnosis of a condition that could be causative of sudden death (such as known coronary artery disease, congestive heart failure or terminal cancer).
17. Use of any prescription medication within 14 days prior to dosing.
18. Use of any over the counter (OTC) medication, including herbal products and vitamins, within the 7 days prior to dosing, except acetaminophen. Up to 3 grams per day of acetaminophen is allowed at the discretion of the Investigator prior to dosing.
19. Use of any drugs or substances known to be significant inhibitors of Cytochrome P450 (CYP) enzymes and/or significant inhibitors or substrates of P-glycoprotein (P-gp) and/or Organic anion transporting polypeptides (OATP) within 14 days prior to the first dose of trial drug.
20. Use of any drugs or substances known to be inducers of CYP enzymes and/or P-gp, including St. John's Wort, within 30 days prior to the first dose of trial drug.
21. Blood donation or significant blood loss (volume >500 ml) within 56 days prior to dosing.
22. Plasma donation within 7 days prior to dosing.
23. Participation in another clinical trial within 30 days prior to dosing.
24. Has been on a significantly abnormal diet during the 4 weeks preceding the first dose of trial medication.
25. Unwilling to remove any artificial nails (e.g. acrylic, gel) or fingernail polish and not use such products for the duration of the trial.
26. History or presence of allergic or adverse response to Listerine breath strips or aspartame.

Additionally, the following exclusion applies only to participants in Part 1, the SAD trial: Is lactose intolerant. - The following food and beverages are not allowed from 72 hours prior to dosing up until the end of the confinement period (discharge from the clinic):

* Xanthine-containing products (e.g. coffee, tea, cola, chocolate)
* Alcohol-containing beverages
* Grapefruit, grapefruit juice, and Seville oranges
* Beverages containing quinine (e.g. tonic, bitter lemon) Medications that are excluded for inclusion into the trial should remain restricted until the end of the confinement period

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events in the Single Ascending Dose (SAD) population | from date of the start of treatment through completion of clinical procedures on Day 126
  Subjects will be monitored for any adverse events from the signing of the consent form until the end-of-study visit. The Investigator or a Sub-Investigator will assess its relationship to the study drug.
Number of Participants with Treatment-Related Adverse Events in the Multiple Ascending Dose (MAD) population | from date of the start of treatment through completion of clinical procedures on Day 168
  Subjects will be monitored for any adverse events from the signing of the consent form until the end-of-study visit. The Investigator or a Sub-Investigator will assess its relationship to the study drug.

SECONDARY OUTCOMES:
Pharmacokinetics, Maximum concentration (Cmax), of TBAJ-587 and metabolites | Day(D)1: 0,0.5,1,1.5,2,3,4,5,6,7,8,10,12,16; D2: 24,28,32,36,40,44; D3: 48,54,60,66; D4: 72,78,84,90; D5: 96,108; D6: 120,132; D7: 144,156; D8: 168; D14: 0.5,1,2,3,4,5,6,7,8,12,16,24; D28: 0.5,1,2,3,4,5,6,7,8,12,16,24,36
  Cmax will be calculated from plasma concentrations of TBAJ-587, M2, M3 and M12
Pharmacokinetics, Time of maximum concentration (Tmax), of TBAJ-587 and metabolites | Day(D)1: 0,0.5,1,1.5,2,3,4,5,6,7,8,10,12,16; D2: 24,28,32,36,40,44; D3: 48,54,60,66; D4: 72,78,84,90; D5: 96,108; D6: 120,132; D7: 144,156; D8: 168; D14: 0.5,1,2,3,4,5,6,7,8,12,16,24; D28: 0.5,1,2,3,4,5,6,7,8,12,16,24,36
  Tmax will be calculated from plasma concentrations of TBAJ-587, M2, M3 and M12
Pharmacokinetics, Area under the concentration-time curve (AUC), of TBAJ-587 and metabolites | Day(D)1: 0,0.5,1,1.5,2,3,4,5,6,7,8,10,12,16; D2: 24,28,32,36,40,44; D3: 48,54,60,66; D4: 72,78,84,90; D5: 96,108; D6: 120,132; D7: 144,156; D8: 168; D14: 0.5,1,2,3,4,5,6,7,8,12,16,24; D28: 0.5,1,2,3,4,5,6,7,8,12,16,24,36
  AUC will be calculated from plasma concentrations of TBAJ-587, M2, M3 and M12
Effect of a high-calorie, high-fat meal on the pharmacokinetics of TBAJ-587 | Day 1: 0, 0.5, 1, 1,5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16; Day 2: 24, 28, 32, 36, 40, 44; Day 3: 48, 54, 60, 66; Day 4: 72, 78, 84, 90; Day 5: 96, 108; Day 6: 120, 132; Day 7: 144, 156; Day 8: 168
  Geometric mean ratio of TBAJ-587's area under the (plasma concentration vs. time) curve when administered with a high-calorie, high-fat meal versus when administered in the fasting state, and similarly for the maximum concentration. Inference will be based on analysis of variance applied to log-transformed parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Bruinenberg, MD, MBA, Study Chair — Global Alliance for TB Drug Development
Locations (1):
- QPS Netherlands B.V., Groningen, Netherlands

REFERENCES:
- [Derived] Leding AAM, Bruinenberg P, Conradie A, Nedelman J, Lombardi A, Hickman D, Simonsson USH. Population pharmacokinetics of TBAJ-587 and its main metabolites-Evaluation of different loading dose strategies and early dose selection. Br J Clin Pharmacol. 2025 Nov 19. doi: 10.1002/bcp.70333. Online ahead of print. PMID 41255184
- [Derived] Komm OD, Tyagi S, Garcia A, Almeida D, Chang Y, Li S-Y, Castillo JR, Converse PJ, Black T, Fotouhi N, Nuermberger EL. Contribution of telacebec to novel drug regimens in a murine tuberculosis model. Antimicrob Agents Chemother. 2025 Jan 31;69(1):e0096224. doi: 10.1128/aac.00962-24. Epub 2024 Dec 9. PMID 39651910